CLINICAL TRIAL: NCT04389827
Title: Global Kidney Patient Trials Network
Acronym: GKPTN
Status: Completed | Type: Observational
Sponsor: The George Institute (Other)
Collaborators: Emerald Clinical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GKPTN2019
Record Dates: First submitted 2020-05-04; First posted 2020-05-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Kidney Diseases
Keywords: Chronic Kidney Disease; Diabetic Nephropathy; Hypertensive Kidney Disease; Glomerulonephritis (GN); Focal Segmental Glomerulosclerosis (FSGS); Membranous Nephropathy; Minimal Change Disease; Immunoglobulin A Nephropathy (IgAN); Glomerulonephritis not otherwise specified; GN; FSGS
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Diabetic Nephropathies; Hypertensive Nephropathy; Glomerulonephritis; Glomerulosclerosis, Focal Segmental; Glomerulonephritis, Membranous; Nephrosis, Lipoid; Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Incident & Prevalent Patients: Incident and prevalent patients diagnosed with a kidney disease at participating centres

SUMMARY:
This is a prospective international multi-centre, observational cohort study of incident and prevalent patients diagnosed with a kidney disease

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of primary kidney disease
2. Regular visits (6-12 monthly) with a physician at a participating site that includes the monitoring of protein in urine and kidney function
3. eGFR > 25 ml/min/1.73m2
4. ≥ 2 to ≥ 80 years of age
5. One of the following laboratory urine parameters within 12 months of screening meeting the values of:

   * Urine Albumin-to-Creatinine Ratio (UACR) > 200 mg/g OR
   * Protein-to-Creatinine Ratio (PCR) > 300 mg/g OR
   * Albumin Excretion Rate (AER) > 200 mg/day OR
   * 24 hour Albumin Excretion > 200 mg/day OR
   * 24 hour Urine Protein Excretion > 300 mg/day
6. Willing and able to sign informed consent
7. Willing to be approached about participation in interventional research studies

Exclusion Criteria:

1. Life-expectancy of less than 6 months
2. Currently receiving renal replacement therapy or planned to start in the next 6 months
3. Planned transplant in the next 6 months
4. Currently participating in a clinical trial involving investigational medicinal product (exception is participation in studies implemented through the GKPTN)

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from units that provide a comprehensive nephrology service
Sampling Method: Non-Probability Sample
Enrollment: 5999 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
estimated Glomerular Filtration Rate (eGFR) | Collected Six-Monthly (minimum)
  Routine results
Albuminuria | Collected Six-Monthly (minimum)
  Routine results

CONTACTS AND LOCATIONS:
Overall Officials: Hiddo Lambers Heerspink, Principal Investigator — The George Institute; Sradha Kotwal, Principal Investigator — The George Institute
Locations (1):
- The George Institute, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
The current plan is that only aggregate data will be shared for research purposes. Individual participant data would only be reviewed in incidental findings and only be discussed with the participant in question.

REFERENCES:
- [Background] Luyckx VA, Tonelli M, Stanifer JW. The global burden of kidney disease and the sustainable development goals. Bull World Health Organ. 2018 Jun 1;96(6):414-422D. doi: 10.2471/BLT.17.206441. Epub 2018 Apr 20. PMID 29904224
- [Background] Tonelli M, Muntner P, Lloyd A, Manns BJ, Klarenbach S, Pannu N, James MT, Hemmelgarn BR; Alberta Kidney Disease Network. Risk of coronary events in people with chronic kidney disease compared with those with diabetes: a population-level cohort study. Lancet. 2012 Sep 1;380(9844):807-14. doi: 10.1016/S0140-6736(12)60572-8. Epub 2012 Jun 19. PMID 22717317
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] McGrogan A, Franssen CF, de Vries CS. The incidence of primary glomerulonephritis worldwide: a systematic review of the literature. Nephrol Dial Transplant. 2011 Feb;26(2):414-30. doi: 10.1093/ndt/gfq665. Epub 2010 Nov 10. PMID 21068142
- [Background] Strippoli GF, Craig JC, Schena FP. The number, quality, and coverage of randomized controlled trials in nephrology. J Am Soc Nephrol. 2004 Feb;15(2):411-9. doi: 10.1097/01.asn.0000100125.21491.46. PMID 14747388
- [Background] Perkovic V, Craig JC, Chailimpamontree W, Fox CS, Garcia-Garcia G, Benghanem Gharbi M, Jardine MJ, Okpechi IG, Pannu N, Stengel B, Tuttle KR, Uhlig K, Levey AS. Action plan for optimizing the design of clinical trials in chronic kidney disease. Kidney Int Suppl (2011). 2017 Oct;7(2):138-144. doi: 10.1016/j.kisu.2017.07.009. Epub 2017 Sep 20. PMID 30675428
- [Background] de Zeeuw D, Heerspink HJL, Jardine M, Perkovic V. Renal trials in diabetes need a platform: time for a global approach? Lancet Diabetes Endocrinol. 2018 May;6(5):356-358. doi: 10.1016/S2213-8587(17)30263-2. Epub 2017 Aug 7. No abstract available. PMID 28797748
- [Background] Woodcock J, LaVange LM. Master Protocols to Study Multiple Therapies, Multiple Diseases, or Both. N Engl J Med. 2017 Jul 6;377(1):62-70. doi: 10.1056/NEJMra1510062. No abstract available. PMID 28679092
- [Background] Berry SM, Connor JT, Lewis RJ. The platform trial: an efficient strategy for evaluating multiple treatments. JAMA. 2015 Apr 28;313(16):1619-20. doi: 10.1001/jama.2015.2316. No abstract available. PMID 25799162
- [Background] Parker CC, James ND, Brawley CD, Clarke NW, Hoyle AP, Ali A, Ritchie AWS, Attard G, Chowdhury S, Cross W, Dearnaley DP, Gillessen S, Gilson C, Jones RJ, Langley RE, Malik ZI, Mason MD, Matheson D, Millman R, Russell JM, Thalmann GN, Amos CL, Alonzi R, Bahl A, Birtle A, Din O, Douis H, Eswar C, Gale J, Gannon MR, Jonnada S, Khaksar S, Lester JF, O'Sullivan JM, Parikh OA, Pedley ID, Pudney DM, Sheehan DJ, Srihari NN, Tran ATH, Parmar MKB, Sydes MR; Systemic Therapy for Advanced or Metastatic Prostate cancer: Evaluation of Drug Efficacy (STAMPEDE) investigators. Radiotherapy to the primary tumour for newly diagnosed, metastatic prostate cancer (STAMPEDE): a randomised controlled phase 3 trial. Lancet. 2018 Dec 1;392(10162):2353-2366. doi: 10.1016/S0140-6736(18)32486-3. Epub 2018 Oct 21. PMID 30355464
- [Background] Park JW, Liu MC, Yee D, Yau C, van 't Veer LJ, Symmans WF, Paoloni M, Perlmutter J, Hylton NM, Hogarth M, DeMichele A, Buxton MB, Chien AJ, Wallace AM, Boughey JC, Haddad TC, Chui SY, Kemmer KA, Kaplan HG, Isaacs C, Nanda R, Tripathy D, Albain KS, Edmiston KK, Elias AD, Northfelt DW, Pusztai L, Moulder SL, Lang JE, Viscusi RK, Euhus DM, Haley BB, Khan QJ, Wood WC, Melisko M, Schwab R, Helsten T, Lyandres J, Davis SE, Hirst GL, Sanil A, Esserman LJ, Berry DA; I-SPY 2 Investigators. Adaptive Randomization of Neratinib in Early Breast Cancer. N Engl J Med. 2016 Jul 7;375(1):11-22. doi: 10.1056/NEJMoa1513750. PMID 27406346
- [Background] Kim ES, Herbst RS, Wistuba II, Lee JJ, Blumenschein GR Jr, Tsao A, Stewart DJ, Hicks ME, Erasmus J Jr, Gupta S, Alden CM, Liu S, Tang X, Khuri FR, Tran HT, Johnson BE, Heymach JV, Mao L, Fossella F, Kies MS, Papadimitrakopoulou V, Davis SE, Lippman SM, Hong WK. The BATTLE trial: personalizing therapy for lung cancer. Cancer Discov. 2011 Jun;1(1):44-53. doi: 10.1158/2159-8274.CD-10-0010. Epub 2011 Jun 1. PMID 22586319
- [Result] Kotwal SS, Perkovic V, Jardine MJ, Kim D, Shah NA, Lin E, Coggan S, Billot L, Vart P, Wheeler DC, de Boer IH, Zhang H, Hou FF, Sugawara Y, Marion J, Lewis RJ, Berry LR, McGlothlin A, Jha V, De Nicola L, Gorriz JL, Heerspink HJL; GKPTN and CAPTIVATE Investigators. The Global Kidney Patient Trials Network and the CAPTIVATE Platform Clinical Trial Design: A Trial Protocol. JAMA Netw Open. 2024 Dec 2;7(12):e2449998. doi: 10.1001/jamanetworkopen.2024.49998. PMID 39661388
- See also: International Diabetes Federation (IDF). IDF Diabetes Atlas 8th edn. Brussels, Belgium:: International Diabetes Federation; 2017 — http://www.diabetesatlas.org